CLINICAL TRIAL: NCT03404856
Title: Study of ORL-1G (D-galactose) in Patients With Glycogen Storage Disease Type 14
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orpha Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GALA-1
Record Dates: First submitted 2018-01-13; First posted 2018-01-19 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Glycogen Storage Disease, Type 14
Keywords: CDG It; CDGIt PHOSPHOGLUCOMUTASE 1 DEFICIENCY PGM1 DEFICIENCY GLYCOGEN STORAGE DISEASE XIV; GSD14 GSD XIV
MeSH Terms: conditions — Glycogen Storage Disease; Glycogen Storage Disease XIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with ORL-1G - D-galactose (Other)
  Interventions: Drug: ORL-1G - D-galactose

INTERVENTIONS:
Drug: ORL-1G - D-galactose — Oral ORL-1G - D-galactose

SUMMARY:
Study of ORL-1G in Patients With Glycogen Storage Disease Type 14

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Glycogen Storage Disease Type 14.
* Less than 18 years old.

Exclusion Criteria:

* Diagnosis of any other disease that is not a manifestation of Glycogen Storage Disease Type 14.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in liver function. | 3 months after treatment starts
  Statistically significant decrease in plasma liver enzyme levels

SECONDARY OUTCOMES:
Improvement in serum transferrin glycosylation pattern. | 30 days after treatment starts
  Decreased serum level of hypoglycosylated transferrin.

CONTACTS AND LOCATIONS:
Locations (1):
- Orpha Labs, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided